CLINICAL TRIAL: NCT03488342
Title: Randomized Clinical Trial of Rives Technique Versus Lichtenstein Repair for Primary Inguinal Hernia
Brief Title: Rives Technique Versus Lichtenstein Repair for Primary Inguinal Hernia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Siberia-Serena (Other)
Responsible Party: Principal Investigator, José Jacob Motos Micó, Principal Investigator, Hospital Siberia-Serena
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HSiberia-Serena
Record Dates: First submitted 2018-03-22; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Primary Inguinal Hernia
Keywords: Rives technique; Lichtenstein repair
MeSH Terms: interventions — Wound Healing

STUDY DESIGN:
Intervention Model Description: randomized,controlled and double-blind study
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rives technique (Other): Rives technique for primary inguinal hernia
  Interventions: Procedure: Repair for primary inguinal hernia
- Lichtenstein repair (Other): Lichtenstein repair for primary inguinal hernia
  Interventions: Procedure: Repair for primary inguinal hernia

INTERVENTIONS:
Procedure: Repair for primary inguinal hernia — Repair for primary inguinal hernia

SUMMARY:
Lichtenstein technique, inserting a mesh over the inguinal cord in the neurological plane, is considered the standard of inguinal hernia repair, but it has 4% recurrence and 12% chronic postoperative pain. Rives technique inserts the mesh in the preperitoneal space behind the neurological plane and the muscular plane, thus better fulfilling the principle of hydrostatics.

DETAILED DESCRIPTION:
These techniques have not been compared randomly for assessment of chronic pain, postoperative complications and recurrences

ELIGIBILITY:
Inclusion Criteria:

Men or women aged between 18 and 93 years (inclusive) at the time of the first screening visit.

They must provide signed written informed consent and agree to comply the study protocol

Exclusion Criteria:

Refusal to give informed consent. Refusal to participate giant inguinal hernias

Ages: 18 Years to 93 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 600 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Evaluate postoperative complications of pain | 7 days
  The patients are clinically reviewed in the office within 7 days of discharge (pain is evaluated at rest and with movement (standing up, sitting down, and walking), using a VAS (visual analogue scale). Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in post- surgical patients, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)

SECONDARY OUTCOMES:
Evaluate the chronic pain | 1 year
  The patients are reviewed clinically by the service's surgeons again after a year. If pain is found, this is evaluated as being with movement, spontaneous, episodic, or constant in nature, and measured with a VAS. The patients are clinically reviewed in the office: pain is evaluated at rest and with movement (standing up, sitting down, and walking), using a VAS (visual analogue scale). Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in post- surgical patients, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)
Evaluate the recurrences | 1 year
  The patients are reviewed clinically by the service's surgeons again after a year. The inguinal region is examined. A mass, reducible or otherwise, is regarded as a recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Siberia Serena, Talarrubias, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: Undecided